## PROMOTING PHYSICAL ACTIVITY IN HIGH POVERTY NEIGHBORHOODS

**Procedures Manual** 

October 2013

This manual was prepared by the project team for use in the project titled Promoting Physical Activity in High Poverty Neighborhoods.

# **TABLE OF CONTENTS**

| Introduction | 4 |
|----------------------------------------|------------------------------|
| Equipment | 5 |
| Apple iPad Mini | 5 |
| Pendragon Forms VI | 5 |
| Park Counters | 5 |
| Equipment Management and Distribution | 5 |
| Data Collection | 5 |
| Participant Recruitment and Protection | 6 |
| Park Use Counters | 6 |
| Installation on an iPad | 7 |
| Counter use | 8 |
| Pendragon Data Entry Forms | 9 |
| Park scan | 9 |
| Survey/Entrevista | 10 |
| Environmental scan | 10 |
| Path scan | 11 |
| Fitness Zone scan | 12 |
| Data Reliability | 13 |
| Target Area Pictures | 13 |
| Image file transfer and storage | 14 |
| File naming protocol | |
| Data Management | 14 |
| Data Protection | 14 |
| Field Logs | 14 |
| Pendragon Forms VI | 14 |
| Initiation | 14 |
| Creating users | 15 |
| Form freezing | 15 |
| Form distribution | 16 |
| Creating groups | 16 |
| Data Sync (iPad to laptop) | 17 |

| | Data Transfer | 18 |
|----|------------------------------------------------------|----|
| | Data export | 18 |
| | Data file upload | 19 |
| ٩р | pendices | 22 |
| | Appendix A: Park counters | 22 |
| | Appendix B: Park mapping guide | 23 |
| | Appendix C: Park user and household survey (English) | 31 |
| | Appendix D: Park user and household survey (Spanish) | 37 |
| | Appendix E: Body type categories | 43 |
| | Appendix F: Park user interview recruitment guide | 44 |
| | Appendix G: Household interview recruitment guide | 46 |
| | Appendix H: Oral consent script | 49 |
| | Appendix I: Project summary (English and Spanish) | 50 |
| | Appendix J: Emergency services information | 52 |
| | Appendix K: Data and safety monitoring plan | 53 |
| | Appendix L: Data Log | 56 |
| | Appendix M: Setting the network IP address | 58 |

#### Introduction

While routine physical activity is critical to optimal health, our preliminary studies have indicated that residents of low-income communities in Los Angeles are less likely to exercise than those in high-income communities, and they are less likely to use their neighborhood parks, even when the parks are within walking distance. Parks in low-income neighborhoods tend to be smaller and serve a greater population density, but even after accounting for the size and the population served, they are still used less than parks in wealthier neighborhoods. In our preliminary studies, we found that parks in low-income neighborhoods also had fewer part-time staff and offered fewer programs and organized activities than parks in higher-income areas, and these factors partly accounted for their lower use. As well, parks in low-income neighborhoods are often perceived as less safe, a characteristic associated with lower use. Simultaneously, the lack of use and dearth of programming may contribute to a perception of lack of safety, creating a vicious cycle. Nonetheless, we have documented that when parks in low-income neighborhoods offer events and activities, they can be just as busy as parks in higher-income areas. We hypothesize that limited park use in low-income areas can be attributed to the lack of organized and reliable infrastructure of activities that meet the needs of local residents and that offering more activities and programs in parks will increase park use and park-based physical activity.

According to the Task Force on Community Level Preventive Services, community-level campaigns are both effective and scalable. For the past eight years, we have conducted research in public neighborhood parks and found that these venues offer great potential for increasing physical activity for populations. Based upon this work, as well as our previous work on the cost-effectiveness of physical activity interventions, we propose to test community-level campaigns targeting low-income populations that will be relatively low-cost and easy to replicate.

The study has three specific aims:

- 1. Using a full factorial design, compare whether park use and population physical activity in low-income neighborhoods increase with the availability of a) more organized physical activity classes, including Zumba, line dancing, and aerobics indoors and outdoors, and/or b) a loyalty program approach that rewards frequent park users.
- 2. Determine whether either of these two approaches changes the perception of park safety and neighborhood safety.
- 3. Identify the cost effectiveness of both approaches in terms of dollars spent to generate increased physical activity in parks as measured through systematic observation.

This manual describes study protocols and instruments specific to this study. The full SOPARC manual is not included here; however, a brief summary of how it is implemented is described in the Data Collection section. Similarly, only the steps in Pendragon Forms VI that necessary for project functioning are described here. The full manual is available for download from the vendor website (http://www.pendragonsoftware.com/).

### **EQUIPMENT**

To accomplish the goals stated above, we will use several different data collection instruments loaded onto a single device. Some of these instruments will be accessed via Pendragon Forms VI, while others are standalone applications developed by RAND for this project. The third party software and hardware used are described briefly below. Each will be discussed in greater detail in later sections describing their use.

## Apple iPad Mini

All data collection instruments will be fielded on this device. These are 16GB, WiFi-enabled (i.e., no data plan) devices. Each Mini includes one USB wall charger. Manuals and other documentation are available online.

These devices are not linked to an iTunes or iCloud account, email account, or calendar. Data collectors should be instructed not to link them to any accounts or access iTunes or iCloud on these devices. RAND has logged each of these devices and has the serial numbers and equipment numbers on file.

## Setup and daily care

These devices are not to be opened in any way, and settings should be managed by the project manager only. Outside of settings that affect immediate use (e.g., brightness, volume) field staff should be instructed not to alter settings to avoid any interruption of Pendragon or the other project applications.

IPads are to be charged the night before use in the field using the Apple charger only. Whenever possible a surge protector should be used.

## **Pendragon Forms VI**

This software allows the user to create custom data collection forms that are output in HTML5 applications that run while disconnected from a network. Data collected on the handhelds are synchronized into Microsoft Access. All data will be entered in one of five forms created in this application.

## **Park Counters**

These applications were developed by RAND specifically for this project, and are standalone counter applications that observers will use to record park utilization. There are two park counters, one records gender, age, and activity level, and one records gender by race/ethnicity. See Appendix A for a screenshot and further description of each counter.

# **Equipment Management and Distribution**

The RAND supplied field laptop (Dell E6410), iPads not in use, and park folders will be stored at AltaMed. Promotoras are to charge their own iPad overnight after conducting park observations, or drop off at AltaMed for charging if they are not scheduled to work in parks.

## **DATA COLLECTION**

The two primary pieces of data collection are park observations and interviews. Observations are conducted according to SOPARC protocols, on three weekdays and three weekend days spread over

five to six months. Observations occur three times per day at 3-hour intervals (e.g., 12pm, 3pm, 6pm). A team of two *promotoras* is assigned to collect data at a park, though at the beginning of the data collection phase two teams of two were assigned for reliability assessment purposes.

Prior to beginning data collection project managers will visit each park and create a target area map (see appendix B for a park mapping guide). On the first day of data collection a project manager meets the team at the park to review the park map and deliver any needed equipment and/or materials. On subsequent data collection days a project manager will meet the team if they have not observed at that park previously, otherwise the team will proceed according to the schedule and data collection protocols.

There are two primary types of interviews; targeted park user interviews (people in the park) and randomly selected residents (people living within one mile of the park). If *promotoras* are unable to contact residents at home for accessibility, safety, or other reasons, station interviews will be conducted. Station interviews are administered to a convenience sample of individuals who are recruited at high pedestrian spots (e.g., transit stations, storefronts, etc.) in neighborhoods within one mile of the park. The same instrument is used for the three types of interviews (see appendices C and D for English and Spanish versions). Data collectors will record an observed body type for each respondent using an image of body type categories (see appendix E).

## **Participant Recruitment and Protection**

In order to obtain random samples, park user and household interview respondents are recruited according to established protocols. Park users are recruited according to set quotas aimed at gaining participants equally distributed by gender, activity level, and age. Household respondents are recruited using a random selection of residential addresses. Recruitment protocols for both interview types can be found in appendices F and G.

Data collectors will obtain oral consent (appendix H) prior to administering the interview, and provide a small incentive upon completion. They also will have available a project summary sheet (in English and Spanish) that lists the project managers contact information if respondents request additional information (appendix I). If a respondent appears in need of immediate mental health services, data collectors will provide contact information for appropriate emergency services (appendix J) and inform park staff.

## **Park Use Counters**

The 12-button age/activity counter app is designed to capture the number of park users by physical activity level and age group, i.e., observers will record physical activity and age group simultaneously for each individual park user within a defined target area. The app is for counting purposes only and the data must be entered into a separate Pendragon form described below.

The counter consists of 12 buttons arranged in four columns (age group) and three rows (activity level). Buttons are color coded by age group.

On the bottom of the app screen are summary and other functions including:

- 1. Observation Count: Returns a summary of the current counts.
- 2. Reset Counters: Returns all fields to a 0 value.
- 3. Edit Previous Record: Allows the observer to edit the immediately preceding entry.

#### Installation on an iPad

These instructions are for an iPad running iOS 7, and may be different for other devices or operating system. Safari was used to load the counters and the bookmarking and icon creation process described here may vary in other browsers.

- 1. Connect the device to a wireless network.
- 2. Open Safari on the device and navigate to http://mmicdata.rand.org/parkcounter.
- 3. Tap the 'Age/Activity' tab.



- 4. After arriving to the counter screen, tap the save icon on the toolbar, and choose "Add to Home Screen." This will install the icon on the home screen.
  - a. At this point you may choose to change the icon label, which will appear on the screen next to the icon. For this project the icon is labeled 'Age / Activity'.



- 5. While still connected to a wireless network, exit the browser and open the counter appusing the icon that you just created to ensure that it loaded properly.
- 6. Exit the counter app and turn off the wireless connection.
- 7. Reopen the counter app while the wireless connection is off to ensure that it will work in offline mode.

#### Counter use

- 1. Confirm that the counter is reset to all 0s before beginning the observation.
  - a. Resetting the counter after each target area will help to avoid mistakes in subsequent target areas.
- 2. Record each individual according to the established SOPARC protocol.
- 3. When the scan is complete, tap the 'Observation Count' tab to view the recorded data.
- 4. Enter the data into a data entry form.
- 5. Tap the 'Reset Counter' tab to erase counts and return all fields to a 0 value.
- 6. Proceed to the next scan.
  - a. The next scan may be a different target area or a different gender, depending on how observations are structured.

The 8-button counter race/ethnicity app is designed to capture the number of park users by gender and race/ethnicity, i.e., observers will record gender and race/ethnicity simultaneously for each individual park user within a defined target area. The app is for counting purposes only and the data must be entered into a separate Pendragon form described below.

The counter consists of eight buttons arranged in four columns (race/ethnicity) and two rows (gender). Buttons are color coded by race/ethnicity.

On the bottom of the app screen you will find the same summary and other functions included in the 12-button counter:

- 1. Observation Count: Returns a summary of the current counts.
- 2. Reset Counters: Returns all fields to a 0 value.
- 3. Edit Previous Record: Allows the observer to edit the immediately preceding entry.

The installation instructions for this counter are the same as described above for the 12-button counter, except for upon arriving to the installation website, tap the 'Gender/Ethnicity' tab.



## **Pendragon Data Entry Forms**

All data will be entered into a Pendragon Form, each of which is described below.

#### Park scan

This form is used to record park observation data. Each park will have a unique park scan form so that observational data is stored in park specific Access tables. These data are not tagged with a park identifier so it is very important that the correct park scan form is used.

The park scan form contains the following data fields.

<u>Date</u>: Check to ensure that the date is correct.

Time: Check to ensure that the time is correct.

Target area: Enter the number of the target area to be scanned.

<u>Subtarget area</u>: Enter the number of the subtarget area to be scanned. For example, if a target area is divided into three subtarget areas, enter a '1' in this blank for the first subtarget area scanned, and a 2 and 3 for the subsequent scans.

<u>Target area conditions</u>: Tap the appropriate Yes No answer box for each of the following seven contextual variables:

- Accessible
  - Equipped
- Organized
- Empty

- Supervised
- Usable
- Dark

<u>Primary Female activity type</u>: Tap the lookup box to choose the appropriate activity.

<u>Check if no females</u>: Check this box only if no females are present in the target area. Checking this box will advance you to the Primary Male activity type screen.

<u>Females SEDENTARY</u>: Enter the number of sedentary females in each of the four age categories. If there are no individuals in a given age group, leave the field blank.

<u>Females MODERATE</u>: Enter the number of moderately active females in each of the four age categories. If there are no individuals in a given age group, leave the field blank.

<u>Females VIGOROUS</u>: Enter the number of vigorously active females in each of the four age categories. If there are no individuals in a given age group, leave the field blank.

<u>Females Race/Ethnicity</u>: Enter the number of females in each of the four race/ethnicity categories. If there are no individuals in a given group, leave the field blank.

Primary Male activity type: Tap the lookup box to choose the appropriate activity.

<u>Check if no males</u>: Check this box if no males are present in the target area. Checking this box will advance you to the final screen.

<u>Males SEDENTARY</u>: Enter the number of sedentary males in each of the four age categories. If there are no individuals in a given age group, leave the field blank.

<u>Males MODERATE</u>: Enter the number of moderately active males in each of the four age categories. If there are no individuals in a given age group, leave the field blank.

<u>Males VIGOROUS</u>: Enter the number of vigorously active males in each of the four age categories. If there are no individuals in a given age group, leave the field blank.

<u>Males Race/Ethnicity</u>: Enter the number of males in each of the four race/ethnicity categories. If there are no individuals in a given group, leave the field blank.

<u>Scan Complete</u>: Check this box at the end of each target area scan. Tap the "End" tab after checking the box.

## Survey/Entrevista

The English and Spanish versions of the survey are separate forms in Pendragon. Interviewers are required to enter the name of the park in which the interview is administered. Therefore, there will be a single Survey form and a single Entrevista form that will be used across all parks.

The full survey is available in the appendices. Highlighted here are some fields that will assist with data management.

<u>Park user activity level</u>: Choose either Active or Sedentary to indicate the level of activity of the park user survey respondent. This field is completed for park user surveys only.

<u>Partial Survey</u>: This check box is located on the final screen of the Survey/Entrevista form. Check this box if you begin a survey, but are unable to complete it for any reason (e.g., participant chooses to end it early). If you complete the full survey leave this box unchecked.

<u>Full survey completed</u>: Check this box if you administer the full survey, even if the participant chooses not to answer some of the questions. If you checked the Partial Survey box, do not check this box.

## Environmental scan

This form is used to provide an overall impression of the park after each park scan is complete (e.g., 3x/day). Only one person from the team needs to enter the data, but team members should discuss the items as needed to come to an accurate assessment.

Observers are required to enter the name of the park being assessed. Therefore, there will be a single Environmental scan form that will be used across all parks.

The environmental scan form contains the following data fields.

<u>Date and Time</u>: Check to ensure that the proper date and time are displayed.

Park name: Choose the appropriate park from the lookup list.

<u>Your name</u>: Choose your name from the lookup list.

Weather: Mark 'Yes' or 'No' for each of the four items listed below:

- Windy
- Pleasant
- Too cold
- Too hot

Safety: Mark 'Yes' or 'No' for each of the four items listed below:

- Conflict (fight)
- Gang members

- Stray dogs
- Intoxicated people
- People smoking
- Intimidating groups of people

<u>Homeless</u>: Choose the appropriate range to indicate the number of homeless persons present in the park during the scan.

<u>Are there food/drink/snack vendors IN the park?</u> Mark 'Yes' or 'No' to indicate whether there are food vendors selling food or drinks inside the park boundaries.

<u>Are there food/drink/snack vendors AROUND the park?</u> Mark 'Yes' or 'No' to indicate whether there are food vendors selling food or drinks outside the park boundaries, but in the adjacent area (e.g., on the surrounding sidewalk).

<u>Is there major construction or maintenance at the park?</u> Mark 'Yes' or 'No' to indicate whether there is significant construction underway that prohibits accessibility to some target areas.

<u>Marketing materials seen in the park</u>: Mark 'Yes' or 'No' to indicate if the items below are seen around the park.

- Banners
- Posters
- Signes

<u>Complete</u>: Check the box to complete the scan.

## Path scan

This form is only created for those parks that have a walking/running path or track that will be observed as a whole, rather than being included in target areas.

The form is designed to be completed once in its entirety for each park user who passes the counting station during the assigned counting period. The observer should open this form as soon as the counting period begins.

Each park that has a walking path/track will have a unique path scan form so that path scan data is stored in park specific Access tables. Path scan data are not tagged with a park identifier so it is very important that the correct path scan form is used.

The path scan form contains the following data fields.

Date: Check to ensure that the correct date is displayed.

Time: Check to ensure that the correct time is displayed.

<u>Check below if no people are observed</u>: Check this box only if no park users passed the counting station during the assigned time period.

 Note: If no persons pass the counting station during the counting period, the observer should not advance past this first screen during the counting period.

Male: Check this box if the person being recorded is male.

Female: Check this box if the person being recorded is female.

<u>Child</u>: Check this box if the person being recorded is aged 0-12 years.

<u>Teen</u>: Check this box if the person being recorded is aged 13-20 years.

Adult: Check this box if the person being recorded is aged 21-59 years.

Senior: Check this box if the person being recorded is aged 60+ years.

Latino: Check this box if the person being recorded is Latino/Hispanic.

<u>Black</u>: Check this box if the person being recorded is black.

White: Check this box if the person being recorded is white.

Other: Check this box if the person being recorded is another race.

<u>Walk</u>: Check this box if the person being recorded is walking when s/he passes the counting station.

Run: Check this box if the person being recorded is running when s/he passes the counting station

<u>Bike</u>: Check this box if the person being recorded is on a bike when s/he passes the counting station.

<u>Skate</u>: Check this box if the person being recorded is skating (e.g., skates, skateboard) when s/he passes the counting station.

<u>Sedentary</u>: Check this box if the person being recorded is sedentary when s/he passes the counting station (e.g., being pushed in a stroller or wheelchair).

END: Check this box after each person is recorded.

#### Fitness Zone scan

This form is created for those parks that have Fitness Zone(s). Parks may have a single Fitness Zone (FZ) or there may be multiple FZs distributed throughout the park or around a walking path. Fitness Zone equipment is often relatively new (since 2009 or so), has moving parts, and is designed such that users will use their own body weight as resistance. Sand areas containing older, non-moving equipment are most often not observed as FZs.

This form is designed to be completed in its entirety for each individual in the FZ space. If there is more than one person using a piece of equipment, the form should be completed for each individual separately. Each piece of equipment is to be observed in the order established on the map, and as ordered in the form.

Each FZ also should have an entry for Other, which is used to record individuals who are in the FZ space but not using the equipment at the moment of observation. Individuals in the FZ but not using equipment are recorded after all FZ equipment has been observed. There should be an entry for Other even if there are no relevant park users to record.

The FZ scan form contains the following data fields.

<u>Date</u>: Check to ensure that the correct date is displayed.

Time: Check to ensure that the correct time is displayed.

<u>Station ID</u>: Choose the appropriate piece of equipment from the drop-down menu. The order in which equipment is listed in the menu should match the order indicated on the park map, and is the order in which each piece of equipment should be observed.

<u>Check below if no people are observed</u>: Check this box if the piece of equipment is not in use at the time of observation.

Male: Check this box if the person being recorded is male.

<u>Female</u>: Check this box if the person being recorded is female.

Child: Check this box if the person being recorded is aged 0-12 years.

Teen: Check this box if the person being recorded is aged 13-20 years.

Adult: Check this box if the person being recorded is aged 21-59 years.

Senior: Check this box if the person being recorded is aged 60+ years.

<u>Latino</u>: Check this box if the person being recorded is Latino/Hispanic.

Black: Check this box if the person being recorded is black.

White: Check this box if the person being recorded is white.

Other: Check this box if the person being recorded is another race.

<u>Sedentary</u>: Check this box if the person being recorded is sedentary at the moment of observation.

<u>Moderate</u>: Check this box if the person being recorded is moderately active at the moment of observation.

<u>Vigorous</u>: Check this box if the person being recorded is vigorously active at the moment of observation.

<u>Is the person using the equipment for exercise</u>: Check this box if the person being observed is using the equipment for exercise rather than play or lounging (e.g., sleeping on the sit up bench). This box should not be checked if a person is resting between sets if s/he appears to have been using it for exercise.

END: Check this box after each person is recorded.

#### **DATA RELIABILITY**

In addition to the ongoing monitoring of data collection by RAND staff, we will conduct two separate measurements of data reliability. At the project beginning two teams of promotoras will collect data side by side to create two complete observation data sets, which will be used to analyze data collector agreement on a select combination of the observed variables. The second and continuous assessment of data reliability will compare pictures of target areas to the data collected. This is explained further below.

## **Target Area Pictures**

Data collectors will take a picture of a single target area during each complete park scan, which will serve as reliability checks of the observation data. The specific target area of which the picture should be taken will change over time, so the park maps will indicate which target area should be photographed. Photos should be taken using the iPad camera from a distance that captures the entire target area, and from which identification of park users is not possible.

Image file transfer and storage

RAND staff will manage the transfer of pictures from the iPads to the laptop...

#### **DATA MANAGEMENT**

#### **Data Protection**

Data collection will adhere to protocols established by the Data Safety Management Board and in agreement with RAND Human Subject Protection Committee. See appendix  $\frac{K}{K}$  for the Data Safety and Management Plan.

## Field Logs

Data collectors will keep a running log of all interviews attempted and administered in order to track progress and allow calculation of a response rate. Paper logs are used for this purpose and are kept in a folder created for each park, which data collectors are to carry with them on all data collection days. Park folders are to be stored at AltaMed when not in use at a park. RAND staff will update folders as needed. See appendix L for the log template.

Data collected on these logs are entered into two spreadsheets stored on the project Teamspace site, and can be used to track progress and calculate refusal rates.

## **Pendragon Forms VI**

#### Initiation

The Pendragon interface was loaded onto each iPad at AltaMed using a dedicated project router and network called Rand Wireless. This network has the static IP address 192.168.1.5. See appendix M for instructions on setting the IP address.

Steps for loading the Pendragon interface are as follow:

- 1. Connect the iPad to a wireless network.
- 2. Open a web browser on the iPad.
- 3. Enter the URL <a href="http://www.192.168.1.5:8080/formsvi.">http://www.192.168.1.5:8080/formsvi.</a>
- 4. Tap the INSTALL/RUN link on the resulting Pendragon Forms screen.
- 5. Tap the 'Setup' tab and enter the username (i.e., name of the promotora to whom the iPad is assigned), and the password "parks."
- 6. Tap 'OK' to return to the Pendragon Forms synchronization page.
- 7. Add this page to the home screen as an icon, and then close the browser.
- 8. While the device is still connected to the internet, open Pendragon Forms using the icon just created in step 7.
- 9. Tap the 'Sync' tab, and if prompted enter the same username and password as in step 5.
  - a. This step is critical as it establishes the connection with the laptop, and stores the forms in the local browser cache allowing them to function in offline mode. The forms will not work offline and data will not sync if this step is skipped.
- 10. Press the 'Launch' tab to return to the main Pendragon Forms screen, where you will see any forms that have been synced.

#### Creating users

Once the appropriate number of licenses have been purchased and loaded into Pendragon, a User name and Password must be assigned to each device. To create a new User click the 'Users' tab in the Pendragon Forms Manger to open the Pendragon Transfer Agent (PTA) dialogue box.



Next, click the 'Create New User' tab in the PTA (see preceding image), which will open fields in which you will enter the New User Name and Password. The user name and password should be the same as those entered above in step 5 of Initiation. Click the 'Add' tab to complete the process. Repeat for all devices.

## Form freezing

Before a form can be fielded it must be frozen, which locks it for editing and creates an Access table in which data will be stored. Once frozen only a limited amount of editing is possible; see the full Pendragon manual for further discussion of this process (the manual is available as a free PDF download from the Pendragon website).

To freeze a form, highlight it in the Pendragon Forms Manger (PFM) and then click the 'Properties' tab to open the Form Properties dialogue box. Next, click the 'Freeze Form design for distribution to handheld and create database' tab. Click 'Yes' when prompted, and 'OK' to complete the freezing process.



## Form distribution

Once frozen, the form can be distributed (i.e., prepared for assignment to a group as described below). To distribute a form simply highlight it in the Form Designs list and click the 'Distribute' tab. Note that if a form is not frozen the 'Distribute' tab will be grayed out indicating that it cannot yet be distributed (as in the image above).

## Creating groups

Pendragon uses Groups to send distributed forms to devices, and sync data from devices back to the database. Devices included in a group will receive all forms that are assigned to the same group during the sync process. This project uses a single group called Parks that contains all forms and all devices. To create a new group, click the 'Groups' tab to open the PTA. Scroll down past where users were created in the preceding step and click the 'Create New Group' tab, which will open a field in which you will enter the group name. Click the 'Add' tab to complete the process.



Once the group has been created you will see the new group listed in the Groups section of the PTA. Click on the newly created group to add users and forms. All users and distributed forms will be available for adding to the group.

## Data Sync (iPad to laptop)

Data will be synced at AltaMed by RAND staff, with the AltaMed promotora supervisor serving as a backup. Data typically will be synced each Friday morning.

The data sync process is as follows:

- 1. Plug in router to power source.
- 2. Connect Ethernet cable from router to the RAND laptop, which will begin to broadcast the Rand Wireless network.
- 3. Connect a device to the Rand Wireless network.
- 4. Open Pendragon Forms on the device.
- 5. Tap the Sync tab, which will begin the data transfer.

Note: if any form revisions/updates are completed prior to the data transfer, distributed forms will be sent to the iPads during this same sync.



## **Data Transfer**

Once all data has been synced from devices to the laptop, it must be exported and transferred to RAND via a secure file sharing service (i.e., Accellion). Access to this site is available on an individual basis.

There are two steps to the data transfer process, which are explained separately below.

## Data export

Pendragon can export data in .xls, .txt, or .csv format. Data are exported one form (i.e., one Access data table) at a time. To export to Excel, which this project does, open Pendragon on the laptop, highlight the form to be exported, and click on the 'To Excel' tab in the PFM.



Data normally will be exported on a weekly basis, for each park that was observed since the preceding data transfer was completed. In addition to the park specific forms, the Entrevista (All Parks), Survey (All Parks), and Environmental scan (All Parks) should be exported.

Resulting data files should be named in a consistent fashion, as shown below.

Survey: Survey\_mmddyy (e.g., Survey\_093013)

Entrevista: Entrevista mmddyy (e.g., Entrevista 093013)

Environmental scan: EnvScan mmddyy (e.g., EnvScan 093013)

Park scan: Park name\_ParkScan\_mmddyy (e.g., Normandie\_ParkScan\_093013)

Path scan: Park name PathScan mmddyy (e.g., MtCarmel PathScan 093013)

FZ equipment scan: Park name\_FZ\_mmddyy (e.g., South\_FZ\_093013)

Once all files have been created they should be zipped and the folder named as "Parksdata\_mmddyy."

If there is any data cleaning to be done, it should be done prior to zipping the final data files. Any adjustments to the data should be made in the database, and only if you are 100% certain of the changes.

### Data file upload

Once exported and zipped as described above data files are to be transferred to RAND via Accellion's secure file sharing site (https://mft1.rand.org/courier/web/1000@/wmLogin.html).

The steps below explain how to transfer data files into your Accellion workspace for RAND Corporation use. For questions or assistance, please contact Stephanie Williamson at swilliam@rand.org.

### Logging in and setting password

1. Open a web browser and go to https://mft1.rand.org.

2. Enter your email address and the "First time password" that was provided in the email invitation you received from RAND. Click Login.



3. As prompted, set a new password. Enter your "first time" password, then the password you want to use in the future. Your password must be at least 6 characters, including a number and an uppercase letter. Click Update Password. When your password is updated, click OK.



4. When your password is updated, click OK.

## Transferring files to your workspace

1. After you log in, click your workspace name (i.e., ParksRCT) in the Send File window that opens.



2. In the window that opens click 'ToRAND'.



the file (i.e., zipped folder) to be uploaded or highlight it and click 'Open'.

- 5. Click 'Add'.
- 6. You will see an upload status bar, and will see the uploaded files in the ToRAND workspace when the upload is complete.

RAND receives automatic alerts when files are added, so no notification of upload is needed.

### **APPENDICES**

## **Appendix A: Park counters**

Counter 1 consists of 12 color coded buttons, and is designed to capture activity level by age group in a single scan.



Counter 2 consists of eight buttons, and is designed to capture gender by race/ethnicity in a single scan. This scan is to be complete after the activity level by age scan.



#### Appendix B: Park mapping guide

Direct observations are made in designated Target Areas (i.e., a distinct, scannable space) that represent all standard locations likely to provide opportunities for park users to be physically active. These areas will be predetermined and identified for observations prior to baseline assessments. A map is created to identify areas and a standard observation order for each park. It is important to establish the Target Area map prior to initiating the observations.

During occasions of high user density, Target Areas can be subdivided into smaller Subtarget Areas (scan spaces) so that more accurate measures can be obtained (e.g., separate groups of people using opposite ends of a soccer field provide observation challenges without separating the areas). Observers use standard court or field markings or other environmental features to determine appropriate Subtarget Areas within each Target Area. Data from these smaller spaces are summed to provide an overall measure for each Target Area.

NOTE: A decision to subdivide a Target Area depends upon (1) the number of park users in the area, and (2) the type of user activity. Fast moving activities with people clustered together and moving in diverse directions (e.g., during soccer) require smaller scan spaces.

The goal of mapping is to divide parks into smaller, observable sections (i.e., Target Areas) so that accurate park user counts can be made according to SOPARC protocols. A well-defined Target Area is one that can be scanned from left to right without encountering visual obstructions. They should be a size that makes it possible county all individuals within the area accurately. Observing parks without clearly mapped Target Areas can result in inconsistent counting and lower quality data.

## Preparation

- 1. Find out if the park or the parks and recreation department has an existing map.
- 2. Print a satellite image of the park from an online mapping site (e.g., Google Earth, Google Maps).
  - a. The print out should show all areas of the park to be included in the observations.
  - b. Keep in mind that the image may be out of date or missing some features. Additionally, tree coverings may obscure some important features of interest. Nonetheless, this satellite image should provide an outline and general layout of the park and be a good place to start.
- 3. Get a feel for the layout of the park and how it is used.
  - a. Take a walk around the park and note the general layout and major features.
  - b. Look around to see if there are obvious sections or dividers that can help to define Target Areas.
  - c. Note which parts of the park are the most and least used.
  - d. Make note of any unique park features that may need to be considered for data collection.

### **Defining Target Areas**

 A target area is a space in which activities may occur. A target area should be large enough to accommodate activity, but small enough to accurately count everyone who may be using the area.

- 2. Areas of the park that generally are open to the public for use should be observed. Areas not intended for public use or that would be inappropriate for observation (e.g., storage space, staff offices, restrooms) should not be included in SOPARC observations.
- 3. There is no established minimum or maximum number of Target Areas, nor is there a defined size limit for a Target Area. Parks with large numbers of Target Areas may require more than one observer working simultaneously.
- 4. Data collectors need to be able to move efficiently from area to area during an observation rotation.
- 5. Data collectors should be able to observe the entire Target Area from one spot on the ground, and be able to scan from left to right without visual obstruction.
- 6. If possible, each Target Area should be made up of one primary feature (e.g., Lawn, Sidewalk, Basketball Court, Play area, Gym, Classroom). This permits the aggregation of data for similar Target Areas within the same park or across parks. However, this may not always be possible, and some areas may have mixed characteristics (e.g., Lawn and Sidewalk).
  - a. When you enter Target Areas with mixed characteristics into the SOPARC online app, name it according to its primary characteristic.
- 7. Existing boundaries (e.g., chalk lines on fields, tree lines, fences) can help determine a Target Area.
  - a. Keep in mind that Target Areas need to remain the same throughout the observation periods and that chalk lines may be temporary and may change from one sport or season to the next.
- 8. Activity types can also be used to help define Target Areas. For example, a tree-shaded section of a large green space could be divided into a separate Target Area since one might expect to observe people having picnics or being involved in some other sedentary activity, rather than running around or playing a sport as in the open space.

### **Ordering Target Areas**

- 1. Order Target Areas such that the data collector can move clockwise through the park efficiently.
- 2. It may be possible to observe multiple Target Areas from a single point order them accordingly.
- 3. By convention, begin observation rotations in the gymnasium, auditorium, community center, or comparable indoor space if there is one.
  - a. If there is no gymnasium, begin observations at the most prominent indoor space (or outdoor if there are no indoor areas).
  - b. If there are no indoor facilities intended for public use, begin with the most prominent outdoor area (e.g., basketball court, baseball or soccer field, picnic area).
- 4. Avoid having data collectors go into dangerous park areas. If these areas are to be observed, do this from a safe distance.

## **Drawing the Map**

These directions assume you have a map printed from a mapping website. If none is available, draw areas of the park by hand, following the same general process outlined below.

- 1. If a park does not have indoor facilities, begin with the most prominent outdoor park feature (e.g., basketball court, soccer field, picnic area).
- 2. Proceed from the first outdoor Target Area in a clockwise fashion and continue to add Target Areas until all of the park area to be observed has been included in a Target Area.
- 3. If the park does have indoor facilities, begin with the main park building. Draw in any targeted indoor areas, as only the exterior of the building will be shown on a satellite image. Indicate all indoor spaces (e.g., classrooms, hallways, lobbies) on the map. As much as possible, they should be ordered in such a way that the data collector can move efficiently through the Target Areas without having to retrace his/her steps.
  - a. When ordering the indoor Target Areas keep in mind the entrances and exits that can be used to reach other Target Areas.
  - b. If a room has more than one entrance, check to see which is most commonly used and accessible.
- 4. Include non-activity areas on the map to help the data collector locate Target Areas. Number the Target Areas, beginning with the gymnasium (or other prominent indoor space if there is no gymnasium).
- 5. When all indoor spaces have been added to the map and numbered exit the building through the main entrance and begin to draw in the outdoor Target Areas. Continue to add Target Areas until all park areas are represented on the map.
- 6. See notes below on how to create Target Areas from common outdoor spaces.
- 7. Landscaped areas are generally not observed as individual Target Areas (except for gardens with paths or that are designed for use).
  - a. Landscaping may be included in other Target Areas. For example, a green space with landscaped borders might be one Target Area.
- 8. If there is a walking path or trail it should be marked on the map as a single Target Area, not divided and included as a part of other Target Areas.
  - a. Refer to the SOPARC manual for instructions on how to observe walking paths and trails.
- 9. Choose a single point from which the walking path will be observed during every observation. It should be unobstructed, shaded if possible, and in a spot from which you will likely see all individuals using the walking path.

Below are notes on common, individual park areas:

## **Lawns and Other Undefined Green Spaces**

People can use green space for diverse purposes (from sleeping to running) and in varying numbers (one to hundreds of people). Since these areas are of mixed use it can be difficult to obtain an accurate count if they are too large. It is generally best to divide them into smaller, more manageable Target Areas, even though they may be vacant frequently.

1. Use natural boundaries to delineate these Target Areas as much as possible.

- 2. In the absence of obvious boundaries (e.g., fence), use trees, bushes, light posts, tables, and other immovable objects to help create boundaries.
  - a. In addition to defining Target Area boundaries, these objects can help a data collector determine where he/she is on the map, but can also clutter the map unnecessarily. Be judicious in what is included on the map.
- 3. If the area is hilly, it may be necessary to further divide it so that the space can be observed without obstruction.
- 4. Use shade to help define Target Areas.
  - a. If one section of a large green space often is shaded and another is not, try to keep them separate as the amount of shade available often affects usage.

#### **Sidewalks**

Sidewalks generally are used for traveling from point A to B. Keeping these areas separate from a typically sedentary area such as a lawn or picnic area will help to more accurately count how many individuals are involved in the primary activity and at what activity level. You may find sidewalks that encircle a play area, basketball court, or other area designed for a specific activity. These sidewalks can be their own Target Area or may be included with the sport or activity specific area. Some things to consider in making this decision is whether a Target Area including the sidewalk would be too large to accurately observe, and whether the sidewalk might be an expected spectator area (remember that spectators only exist during organized activities, so this most often would not apply to play areas).

- 1. Decide if there is a route that often is used as a walking or jogging path. If so, consider doing a walking path scan for this Target Area.
  - a. If you choose to do a walking path observation using sidewalks as the walking path, do not include these sidewalks as additional Target Areas.
- 2. As sidewalks are normally well-defined, simply divide them into manageable sections so that they can be observed accurately.
- 3. When deciding how much of a sidewalk to include in a Target Area, keep in mind that people often will be moving in two different directions.

## **Play Areas**

These areas are usually well-defined, so unless they are unusually large or have structures that obstruct vision keep them as a single area. It can be helpful to identify markers (e.g., lampposts, benches) so that data collectors can create Subtarget Areas on the fly if needed.

## **Sport Related Courts and Spaces**

Mapping a sport related court or space depends largely on the size and kind of court. Unless separated visually, multiple tennis courts potentially can be grouped together as one Target Area as not many individuals play at one time. Unless they are rarely used, neighboring basketball or volleyball courts usually should not be combined, as they may involve many more people and vigorous activity levels than can be easily counted.

## **Sport and Multi-use Fields**

As the name suggests, multi-use fields might be used for soccer, baseball, football, and other activities. Depending on the season, a multi-use field might be lined for a different sport or activity, and these chalk lines can be used to help determine Target Areas. Check with park staff to see if the lines are likely to remain in place throughout the planned observation period.

- 1. Individual baseball fields often can be left intact as there are usually only a few individuals moving at any one time during a game.
  - a. Bleachers can be included as part of the baseball field Target Area or observed separately. If bleachers are included, individuals in the bleachers watching an organized game would be counted as spectators.
- If a park has numerous sport facilities neighboring one another that might all be in use simultaneously during tournaments or other larger organized activities, each field or court should be an individual Target Area, and the map should indicate where Subtarget Areas are likely to be made.
- 3. Soccer or football fields may be divided in halves to make them easier to count, or they can be left whole but with instructions and markers for division into Subtarget Areas as needed.
- 4. It is not uncommon to see soccer played on baseball fields and vice versa. So keep in mind the season during which you will be observing as this may affect how the area should be defined.
- 5. Areas surrounding fields may contain benches or grass that is often used by spectators. Before beginning to observe the park, determine which part of a Target Area is considered the spectator area (remembering that by definition spectators only exist during an organized activity).

### **Finalizing the Map**

When the park map has been drawn, you may choose to create a digital copy using common software that allows you to use shapes to create or add to images, such as Microsoft PowerPoint. Other, more sophisticated mapping software is also available if desired. A computer generated map is not necessary, but may be helpful as it will likely be clearer and easier to read. The images below show three different methods of creating a park map starting with a satellite image of a park.

# Satellite image of a park printed from online mapping tool



SOPARC map created using Microsoft PowerPoint



# Satellite image of a park printed from online mapping tool



SOPARC map using shapes overlaid on a satellite image



# Satellite image of a park printed from online mapping tool



Hand-drawn SOPARC map



□ > 1 hour, but < 2 hours</p>

□ In the past 6 months

□ Between 6 - 11 months ago □ Between 1 - 2 years ago ☐ More than 2 years ago

(Check one)

□ Today

□ This month

6. When was the first time you came to this park?

Revised 6/11/13

#### NEIGHBORHOOD PARKS AM / PM (Circle one) Time: Date: ☐ ¼ mile resident ☐ ½ mile resident □ 1 mile resident Participant type: □ Park user ☐ Station ¼ mile ☐ Station ½ mile ☐ Station 1 mile Activity level: ☐ Sedentary ☐ Active □ Male ☐ Female Age: INTERVIEWER TO READ STATEMENT: This survey is mainly about \_\_\_\_\_\_\_ [park name]. Please think about this park when you answer the questions. How many children under the age of 18 do you have? 2. How do you describe yourself in terms of race or ethnicity? (Check one) (insert number) □ Latino Asian / Pacific Islander □ American Indian / Alaska Native □ White □ Black □ Other \_\_\_\_ 3. How often do you come to this park? (Check one) 7. How do you usually get to the park? (Check one) □ Daily □ Walk □ A few times a week □ Bike □ Once per week □ Car □ A couple times per month Bus or other public transportation ■ Monthly □ Other □ A few times a year □ This is the first time □ Never [skip to #10] 8. What do you usually do while at this park? (Check all that apply) 4. How many times did you visit this park within the past □ Aerobics ☐ Meet friends SEVEN days? □ Baseball/softball □ Playground (insert number) ☐ Sitting in park □ Basketball (indoors) ☐ Don't know □ Basketball (outdoors) ☐ Skating □ Celebrations or picnics □ Soccer 5. On a typical day when you go to the park, how long do □ Classes □ Swimming you stay there? □ Frisbee □ Tennis (Check one) □ Gymnasium activity □ Volleyball O-30 minutes □ 2-3 hours ☐ Gymnastics equipment □ Walking 31-60 minutes >3 hours ☐ Handball □ Walking with dog

9. When you are at this park, do you run into people you know? (Check one) Yes, often □ Rarely

□ Other \_\_\_\_

☐ Yes, sometimes □ No, not at all

| | | 4 | | 1 | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 10. | | u do not visit this | • | | 16. | | crime rate in this neighbor | 1000 | makes it u | nsar | e to |
| | | | | e respondent answered | l | _ | n walks at night. Do you | | | | |
| | Nev | er" to question 3) | | | l | | Strongly agree | | | | |
| | | | | | l | | Agree | | | | |
| | | | | | l | | Disagree | | | | |
| | | | | | l | | Strongly disagree | | | | |
| 11. | | | | park staff with respect to | l | | | | | | |
| | | | ndlin | ess, and professionalism? | l | | | | | | |
| | • | ck one) | _ | _ | 17. | How | often do you go to other p | arks? | (Check on | e) | |
| | | | | _ | l | | Daily | | | | |
| | | В | | | l | | A few times a week | | | | |
| | | С | | Don't know the staff | l | | Once per week | | | | |
| | | | | | l | | A couple of times per mor | ıth | | | |
| | In | nami hawanta d | | u fool the mark in? | l | | Monthly | | | | |
| 12. | | <u>ck one)</u> | o yo | u feel the park is? | l | | A few times a year | | | | |
| | • | • | | | l | | Never | | | | |
| | | Very safe | | | l | _ | Herei | | | | |
| | | Safe | | | l | | | | | | |
| | | Not very safe | | | 18. | Whi | ch of the programs and eve | nts of | ffered at | | |
| | | Not safe at all | | | l | | [park name] are yo | u awa | are of? (Ch | eck ( | all |
| | | | | ring (Short and | l | that | apply) | | | | |
| 13. | | | | rcise? (Check one) | l | | Aerobics or fitness classes | | | | |
| | | I don't usually ex | erci | se . | l | | After school program | | | | |
| | | Park | | | l | | Arts or crafts | | | | |
| | | Home | | | l | | Dance | | | | |
| | | Private health cl | ub | | l | | Holiday events | | | | |
| | | Streets and sides | walk | 5 | l | | Martial arts | | | | |
| | | Other | | | l | П | Senior classes | | | | |
| | | | | | l | | Sports programs or league | ıc | | | |
| | | | | | l | | Other | | | | |
| | | | | | l | | | | | | |
| | | | | agree or disagree with the | l | ш | None | | | | |
| tolle | | • | the | neighborhood surrounding | l | | | | | | |
| | _ | park. | | | l | | | | | | |
| | | | | | 19. | How | do you usually find out ab | out th | ne progran | ns an | ıd |
| | | | | | l | ever | nts that are offered at this p | ark? | | | |
| 14. | Ther | e is a high crime r | ate i | in this neighborhood. Do | l | (Ask | about each individually) | | | | |
| | vou. | _ | | | l | Do | n't find out about programs | (skip | to 20) | | |
| | • | Strongly agree | | | l | Bar | nners | | Yes | | No |
| | _ | Agree | | | l | Em | ail | | Yes | | No |
| | _ | _ | | | l | Flv | ers at park | | Yes | | No |
| | | Disagree | | | l | | ers from child's school | п | Yes | п | No |
| | ш | Strongly disagree | 2 | | l | | m park office | _ | Yes | | No |
| | | | | | I | | | | | | |
| 15. | The | crime rate in this | neig | hborhood makes it unsafe to | I | | iling | _ | Yes | | No |
| | | n walks during the | _ | | I | | ssage/bulletin board | | Yes | _ | No |
| | | Strongly agree | | , | I | | k/RAP website | | Yes | | No |
| | _ | | | | I | | ord of mouth | | Yes | | No |
| | _ | Agree | | | I | | Other | | | | |
| | | Disagree<br>Strongly disagree | | | I | | | | | | |
| | | ATTOROGIST SUCTORS | | | | | | | | | |

| 20. Have you ever participated in a program sponsored at this park? (Check one) Yes No [skip to 23] 21. When was the last time you participated in a program at [park name]? (Check one) Today In the past month In the past 6 months Between 6-11 months ago Between 1-2 years ago | INTERVIEWER TO READ: Because we know that park use can be affected by whether you work, your health, and your exercise habits, we have a few questions about those. Please remember that your answers are anonymous. 26. Are you currently: (Check all that apply) Working full-time Working part-time Self-employed Unemployed, looking for work Retired Disabled |
|---|---|
| ☐ More than 2 years ago | ☐ A student (full or part time) ☐ A stay-at-home parent |
| | □ Other |
| 22. In which programs have you participated within the past twelve months? | |
| Adult sport league | 27. What is your highest level of education completed? |
| Dance classes | (NOTE: If respondent attended school outside of the U.S.<br>indicate the closest equivalent) (Check one) |
| Fitness / aerobics class □ Yes □ No | 6 <sup>th</sup> grade or less |
| Organized walks / hikes | □ 7 <sup>th</sup> -11 <sup>th</sup> grade |
| Park events (e.g., fair) ☐ Yes ☐ No | ☐ High school graduate or GED |
| □ Other | ☐ Some college (but no degree) |
| | □ Associate's degree (AA) |
| | ☐ Bachelor's degree (BA, BS) |
| 23. What is the nearest intersection to your home? | ☐ Some graduate school or graduate degree |
| (INTERVIEWER NOTE: Please indicate complete street | |
| name (i.e., 49 <sup>th</sup> Place or 49 <sup>th</sup> Street). Also verify that | 30. How many times not work do you oppose in physical |
| these streets intersect!) | <ol> <li>How many times per week do you engage in physical<br/>activities such as walking, cycling or any activity that</li> </ol> |
| Major Street | causes increased breathing or heart rate, leg fatigue, or |
| | causes you to perspire? |
| Cross Street | □ 0 [skip to 30] □ 5 |
| | □ 1 □ 6 |
| | □ 2 □ 7 or more |
| 24. Using the map provided, indicate in which buffer the | □ 3 □ Don't know |
| respondent's home is located. | □ 4 |
| □ 0−¼ mile □ ½-1 mile | 29. What is the usual length of these physical activities? |
| ☐ ¼-½ mile ☐ 1+ miles | (Check one) |
| | ☐ Less than 5 minutes |
| | □ > 5, but < 15 minutes |
| 25. How long have you lived at your current address? | ☐ 15-30 minutes |
| (Check one) | □ > 30, but < 45 minutes |
| Less than 1 year | ☐ More than 45 minutes |
| □ 1-2 years | 30. Do you engage in physical activities as part of your work |
| □ > 2 years, but < 5 years □ Between 5 - 9 years | on a regular basis? (Check one) |
| □ 10 years or more | ☐ Yes ☐ No |

| 31. How much time outside of work do you spend watching | | | | | | dso depressed nothing could cheer you up? Would |
|---|---|---|---|---|---|---|
| | television, DVDs or videos, play | | | | you say | |
| | using a computer on an average | day? | (Check | (one) | ☐ All of the time ☐ A little of the time | |
| | □ 0 - 60 minutes | | | | ☐ Most of the time ☐ None of the time | |
| | □ > 1 hour, but < 2 hours | | | | | ☐ Some of the time |
| | □ Between 2 and 4 hours | | | | | |
| | □ > 4 hours, but < 5 hours | | | | | abot |
| | □ 5 hours or more | | | | | ethat everything was an effort? Would you say □ All of the time □ A little of the time |
| | ☐ I don't know | | | | | ☐ Most of the time ☐ None of the time |
| 37 | In general, would you say your | health | ie- | | | ☐ Some of the time |
| 32. | (Check one) | ilcaitii | 13. | | | |
| | ☐ Excellent | | | | | fworthless? Would you say |
| | ☐ Very good | | | | | ☐ All of the time ☐ A little of the time |
| | □ Good | | | | | ☐ Most of the time ☐ None of the time |
| | ☐ Fair | | | | | ☐ Some of the time |
| | □ Poor | | | | | |
| 33. | Has a doctor ever told you that | you ha | eve an | y of t | he | 35. Now thinking about your physical health, which includes |
| | following conditions? | | | | | physical illness and injury, for how many days during the past |
| | Asthma | | Yes | | No | 30 days was your physical health not good? |
| | Diabetes | | Yes | | No | (insert a number 0-30) |
| | High cholesterol | | Yes | | No | |
| | Heart disease | | Yes | | No | |
| | Hypertension | | Yes | | No | 36. What is your height and weight? |
| | Weight problem | | Yes | | No | (INTERVIEWER NOTE: Remind respondent that the survey |
| | | | | | | is anonymous) |
| 34. | The following questions ask abo<br>feeling during the past 30 days. | | • | | | Height — Feet Inches |
| | please tell me whether you hav | | • | | | Meters Centimeters |
| | the time, Most of the time, A lit | | | | | |
| | of the time." | | | | | Weight Pounds |
| | (Check one for each of the 6 que. | stions) | | | | weight |
| | a name of the state of the stat | | | | | Kilograms |
| | anervous? Would you say | | a lissla | of th | e time | |
| | ☐ Most of the time | ш | None o | or the | time | Now I'm going to read some questions about things that |
| | ☐ Some of the time | | | | | people in this park may or may not do. |
| | | | | | | 33 5 |
| | bhopeless? Would you say | <b>y</b> | | | | <ol> <li>For each of these statements, please tell me whether<br/>you strongly agree, agree, disagree, or strongly</li> </ol> |
| | ☐ All of the time | | A little | of th | e time | disagree. |
| | ☐ Most of the time | | None o | of the | time | |
| | ☐ Some of the time | | | | | <ul> <li>People around here are willing to help each other.</li> </ul> |
| | | | | | | ☐ Strongly agree |
| | | | | | | ☐ Agree |
| | crestless or fidgety? Woul | | | | | ☐ Neither agree nor disagree |
| | ☐ All of the time | | | | e time | □ Disagree |
| | ☐ Most of the time | ш | None o | of the | time | ☐ Strongly disagree |
| | ☐ Some of the time | | | | | I |

| | _ | | | |
|---|---|---|---|---|
| | b. | People in this park can be trusted. | INTERVIEWER TO READ: We are planning to develop som | |
| | | ☐ Strongly agree | new prog | grams for the community and the next questions ask |
| | | ☐ Agree | for your | input on these programs. |
| | | ☐ Neither agree nor disagree | | |
| | | □ Disagree | | |
| | | ☐ Strongly disagree | | ou could get a small prize for going to the park, |
| | | | | ch would you prefer? |
| | | | | Water bottle |
| | c. | People in this park generally don't get along with | | Lip balm |
| | | each other. | | Ball |
| | | ☐ Strongly agree | | Frisbee |
| | | □ Agree | | iTunes gift card |
| | | ☐ Neither agree nor disagree | | Other |
| | | □ Disagree | | |
| | | ☐ Strongly disagree | | |
| | | | | e prize was an entry into a lottery for a larger item, |
| | | | whic | ch prize would you like to win? (Check one) |
| | d. | People in this park do not share the same values. | | iPod |
| | | ☐ Strongly agree | | Tablet computer |
| | | □Agree | | \$200 gift card |
| | | ☐ Neither agree nor disagree | | Other |
| | | □ Disagree | | |
| | | ☐ Strongly disagree | | |
| | | | | at exercise classes would you participate in if they |
| | | | l | e offered at this park? (Check all that apply) |
| 38. | For e | ach of the following, please tell me if it is very | | Aerobics |
| | likely, likely, unlikely, or very unlikely that people in this | | | Boot camp |
| | park | would act in the following manner. | | Hip hop dance |
| | _ | | | Line dance |
| | Peop | le in the park would intervene if: | | Kickboxing |
| | a. | Children were spray-painting graffiti | | Pilates |
| | ۵. | | | Salsa |
| | | □ Very likely | | Walking club |
| | | Likely | | Yoga |
| | | ☐ Neither likely nor unlikely | | Zumba |
| | | ☐ Unlikely | | Other |
| | | □ Very unlikely | | |
| | b. | A fight broke out in the park | | ing the WEEK, when would be the best time for you |
| | | □ Very likely | _ | articipate in these classes? |
| | | □ Likely | | Morning (7-10) |
| | | ☐ Neither likely nor unlikely | | Midday (10-1) |
| | | □ Unlikely | 1 | Afternoon (1-5) |
| | | □ Very unlikely | | Evening (5-8)<br>Night (after 8) |
| | | • | | Hight (after 6) |
| | | | 1 | |

| 43. | | to participate in these classes? | this park? |
|---|---|---|---|
| | you | Morning (7-10) | uis park: |
| | | Midday (10-1) | |
| | | Afternoon (1-5) | |
| | | Evening (5-8) | |
| | | Night (after 8) | |
| | | | This is the end of the questionnaire, thank you for participating. |
| | | | 1 |
| 45. | Afte | r the survey is complete, enter the letter (A – J) that co | rresponds to the respondent's body type from the list below. |
| | | (Enter a letter A – J) | |
# Appendix D: Park user and household survey (Spanish)

Revised 6/11/13

| | PARQUES DE VECINDARIO | | | | | | |
|---|---|---|---|---|---|---|---|
| Ent | trevistador Fecha: | | | Hora | : | A | M / PM (Marque una) |
| Tip | o de participante: | a ¼ de m<br>illa statio | | | a ½ milla<br>lla station | | ☐ Vive a 1 milla<br>☐ 1 milla station |
| Sex | xo: | | | Ac | tividad: [ | □ Sed | dentario 🗆 Activo |
| | UNCIADO PARA QUE EL ENTREVISTADOR LO LEA: Esta encues<br>rque]. Piense en este parque al responder a las preguntas. | ta se refi | ere pr | incipalmente | | | [nombre del |
| 1. | ¿Cuántos hijos tiene que tengan menos de 18<br>años? | | | escribiría ust<br>1? (Marque u | | mo e | n términos de raza o |
| | (escriba el número) | | l Lat<br>l Bla<br>l Mo | nco | | estado | s islas del Pacifico<br>ounidense o nativo |
| 3. | uno) Todos los días Varias veces por semana Una vez por semana Un par de veces al mes | 7. | 0 | aalmente cón<br>A pie<br>En bicicleta<br>En auto<br>Bus u otro tr<br>Otro | ransporte p | úblico | |
| | ☐ Una vez al mes ☐ Varias veces al año ☐ Esta es la primera vez ☐ Nunca [pase a #10] | 8. | ¿Qu | é hace por lo<br>rque todas qu | general en | este | parque? |
| 4. | ¿Cuántas veces fue a este parque en los últimos SIETE días? (escriba el número) □ No sabe | | 0 | Aeróbicos<br>Béisbol o sofi<br>Básquetbol (:<br>Básquetbol (: | adentro) | | Encontrarme con<br>amigos<br>Jugar en el área de<br>recreo |
| 5. | En un día normal, cuando va al parque, ¿cuánto tiempo se queda allí? (Marque una) Menos de 30 minutos Entre 2 y 3 horas Entre 31 y 60 minutos 3 horas o más > 1 hora, pero < 2 horas | | _<br>_<br>_ | Celebracione<br>Clases<br>Frisbee<br>Una actividad<br>gimnasio<br>Usar el equip | s o picnics | 0 | Sentarme y relajarme<br>Patinar<br>Fútbol<br>Nadar<br>Tenis<br>Voleibol |
| 6. | ¿Cuándo fue la primera vez que Ud. visitó a este<br>parque? (Marque una)<br>Hoy | | | gimnasia<br>Balonmano<br>Otra | | | Caminar<br>Caminar con el perro |
| | ☐ Este mes ☐ En los últimos 6 meses ☐ Hace > 6 meses, pero < 11 meses ☐ Hace > 1 año, pero < 2 años ☐ Hace más de 2 años | | | | | | |

1

| | | ndo está en el parqu<br>conoce? <i>(Marque u</i> | | ntra con personas | | pelig | do a la tasa de criminal<br>groso salir a caminar por<br>d está | | | | es |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Sí, muy seguido | | Casi nunca | l ' | | | | | | |
| | | Sí, a veces | | Nunca | l | | Muy de acuerdo | | En desacue | rdo | |
| | | | | | | | De acuerdo | | Muy en des | acuero | lo |
| | (solo | o va a este parque, è<br>o pregunta esta preg<br>nca" al número 3) | | sona contestó | 17. | ¿Que | é tan seguido va a otros | parqu | ues? (Marqu | e una) | ) |
| | | | | | l | | Todos los días | | | | |
| | | | | | l | | Varias veces por semar | ıa | | | |
| | | ISE | | | l | | Una vez por semana | | | | |
| | | no calificaría al pers | | onalismo? (Marque | l | | Un par de veces al mes | | | | |
| | una) | • | au, y profesi | onansmo: (wurque | l | | Una vez al mes | | | | |
| | | | | | l | | Varias veces al año | | | | |
| | | A [ | ] D | | l | | Nunca | | | | |
| | | В | ] F | | l | _ | | | | | |
| | | c E | No conoz | co al personal | | | | | | | |
| | | érminos generales, (<br>ue? (Marque una) | qué tan segi | uro le parece el | | | iles de los programas y<br>inbre del parque] conoce | | os ofrecidos | en | _ |
| | | Muy seguro | ☐ No muy | _ | l | | Clases de ejercicio o ae | róbico | os | | |
| | | Seguro | □ Nada se | eguro | l | | Después de escuela | | | | |
| | | | | | l | | Arte | | | | |
| 13. | čNor | rmalmente dónde h | ace ejercicio | ? (Marque una) | l | | Baile | | | | |
| | | No hago ejercicio n | ormalmente | | l | | Eventos festivos | | | | |
| | | En el parque | | | l | | Artes marciales | | | | |
| | | En casa | | | l | | Actividades para tercer | a eda | d | | |
| | | En un gimnasio pri | /ado | | l | | Ligas deportivas | | | | |
| | | En las calles o vere | das | | l | | Otro | | | | |
| | | En otra | | | l | | Ninguno | | | | |
| | _ | | | | l | _ | MILEGIO | | | | |
| decl | araci | qué tan de acuerdo<br>ones sobre el vecin<br>sa de criminalidad ( | dario que ro | dea al | | se of | no se entera usted de lo<br>frecen en este parque?<br>espondan) | | | | que |
| | | a? Usted está | r este veuli | auno es andi (Que | | No | me entero de los progra | amas ( | pase a 20) | | |
| | • | | _ | | Ι. | Bar | ndera | | □ Sí | | No |
| | | Muy de acuerdo | | desacuerdo | | Por | email | | □ sí | | No |
| | | De acuerdo | □ Ми | ıy en desacuerdo | | Vol | antes en el parque | | □ sí | | No |
| | | | | | | Vol | antes en la escuela | | □ sí | | No |
| | | | | | l ' | De | la oficina | | □ sí | | No |
| 15. | Debi | do a la tasa de crim | inalidad de e | ste vecindario. es | | Un | anuncio por correo | | □ sí | | No |
| | | roso salir a caminar | | | l ' | Tab | lón de anuncios | | □ sí | | No |
| | Uste | d está | | | | Pás | ina de web/Internet | | □ sí | | No |
| | п | Muy de acuerdo | □ Fn | desacuerdo | ' | | escuchó de otra persona | | □ sí | | No |
| | | De acuerdo | | ıv en desacuerdo | | | Otra | | | Ī | |
| | | De acuerdo | ⊔ М | ry en desacuerdo | l ' | | | | | | |

| 20. ¿Alguna vez ha participado usted en un programa patrocinado en [nombre del parque]? (Marque una) Sí | 26. ¿Cuál es su situación laboral actual? (Marque todas que correspondan) Trabaja tiempo completo Trabaja tiempo parcial Trabaja por cuenta propia Desempleado, buscando trabajo Jubilado Descapacitado Estudiante Ama de casa Otra |
|---|---|
| ☐ Hace 1 a 2 años ☐ Hace más de 2 años | 27. ¿Cuál es el grado o nivel escolar <u>más alto</u> que ha<br><u>completado</u> ? (Si se educó fuera de los Estados Unidos,<br>marque el equivalente en los Estados Unidos). |
| 22. ¿En qué programas ha participado en los últimos doce meses? | (Marque una sola respuesta) 6º grado o menos (escuela primaria) |
| Liga deportiva para adultos 🔲 Sí 🗆 No | ☐ Entre 7º y 11º grado<br>☐ Se graduó de la secundaria o preparatoria o |
| Clases de baile Sí No Clases de ejercicio o aeróbicos Sí No | equivalencia |
| Clases de ejercicio o aeróbicos 🗆 Sí 🗆 No Caminatas organizadas 🗆 Sí 🗆 No | ☐ Algunos cursos universitarios pero sin título |
| Eventos del parque (una feria) | ☐ Diploma universitario por una carrera de 2 años |
| Otra | ☐ Diploma universitario por una carrera de 4 años |
| | <ul> <li>Algunos cursos de posgrado o recibió un título de<br/>posgrado</li> </ul> |
| 23. ¿Cuáles son las calles más cercanas a su casa que se | |
| cruzan? (Indicar el nombre entero) | 28. ¿Cuántas veces por semana realiza actividades físicas como caminar, montar en bicicleta o alguna otra |
| Calle principal: | actividad que aumente la frecuencia respiratoria o |
| Calle que la cruza: | cardíaca, le canse las piernas o le haga sudar? |
| | □ 0 [pase al 30] □ 5 |
| 24. En el mapa que se le ha dado, indique en qué zona de | □ 1 □ 6 |
| amortiguamiento está situada la casa del entrevistado. | □ 2 □ 7 o más |
| □ 0−¼ milla □ ½-1 milla | □ 3 □ No sabe |
| ☐ ¼-½ milla ☐ 1+ millas | □ 4 |
| 25. ¿Cuánto tiempo ha vivido en su domicilio actual?<br>(Marque una) | |
| ☐ Menos de 1 año ☐ Entre 5 y 9 años ☐ Entre 1 y 2 años ☐ 10 años o más | <ol> <li>¿Cuál es el tiempo usual que pasa haciendo estas<br/>actividades físicas? (Marque una)</li> </ol> |
| □ > 2 años, pero < 5 años | ☐ Menos de 5 minutos ☐ > 30, pero < 45 |
| | □ > 5, pero < 15 minutos □ > 45 minutos |
| PARA QUE EL ENTREVISTADOR LEA: Como sabemos que la | ☐ Entre 15 y 30 minutos |
| frecuencia con la que usted vaya al parque puede depender | |
| de si trabaja, de su salud y de sus hábitos de ejercicio, | |
| tenemos unas pocas preguntas sobre estos temas. Recuerde<br>que sus respuestas son anónimas. | |
| que sus respuestas son anominas. | 1 |

| 30. | ¿Hace ejercicio físico a | | omo | parte ( | de su | 1 | | c. | Inqu | uieto(a) o intranquilo(a | )? Diría | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | trabajo? (Marque una) | ) | | | | | | | | Siempre | | Casi nunca |
| | □ sí | I | <b>-</b> 1 | lo | | | | | | Casi siempre | | Nunca |
| | | | | | | | | | | A veces | | |
| 31. | En un día promedio y f | | | | | | | d. | Tan | deprimido(a) que nada | a podía | animarle? Diría |
| | ¿cuánto tiempo pasa u<br>videos, jugando juegos | | | | | DO | | | п | Siempre | _ | Casi nunca |
| | computadora? (Marqu | | 0 000 | nuo ui | | | | | | Casi siempre | | Nunca |
| | | | | | | | | | | A veces | _ | Nunca |
| | ☐ Entre 0 y 60 minu | | | | | | | | _ | | | |
| | □ >1 hora, pero < 2 □ Entre 2 horas y 4 | | | | | | | e. | Que | todo le suponía un gra | ın esfu | erzo? Diría |
| | □ >4 horas, pero < | | | | | | | | | Siempre | | Casi nunca |
| | ☐ 5 horas o más | 3 110103 | | | | | | | | Casi siempre | | Nunca |
| | □ No sé | | | | | | | | | A veces | | |
| | L 11032 | | | | | | | | | 22 mil ( | | |
| 32. | En términos generales, | ¿cómo ca | lifica | ría su s | alud | , | | f. | Inut | til? Diría | | |
| - | (Marque una) | , ccomo ca | | | - | - | | | | Siempre | | Casi nunca |
| | | | | | | | | | | Casi siempre | | Nunca |
| | | ☐ Regular<br>☐ Mala | | | | | | | | A veces | | |
| | ☐ Muy buena<br>☐ Buena | ⊔ Maia | | | | | 35 | | hora nic | ense en su salud física, | incluid | ac lac |
| | ⊔ buena | | | | | | 1 - | | | dades físicas y las lesio | | |
| | | | | | | | | | | en cuántos de los últir | | |
| 33. | ¿Alguna vez le ha dicho | | • | | ifre ( | de una | | de | e buena | salud física? | | |
| | o más de las condicion | es nombra | | | | | | | | (escriba un númer | n ontre | 0 4 201 |
| | Asma | | | | | No | | _ | | (escriba un numer | o enu e | : U y 3U) |
| | Diabetes | | | | | No | | | | | | |
| | Colesterol aumentado | | | | | No | 36 | | | on su talla y su peso? | | _ |
| | Una enfermedad card | liaca | _ | | | No | | | | ARA EL ENTREVISTADOR | | |
| | Hipertensión | | | | | | | er | ntrevisto | ado que la encuesta es o | ınonım | ia.) |
| | Un problema del peso | ) | | Si | | No | | | _ | pies | D | ulgadas |
| | | | | | | | | 1 | Talla - | | | entímetros |
| 34. | Las siguientes pregunta | as se refier | ren a | cómo : | se ha | 1 | | | - | metros | | enumeuros |
| | sentido en los últimos | 30 días. En | cad | a pregu | ınta | | | | | | | |
| | favor dígame si se ha s | | | | asi | | | | Peso - | libras | | |
| | siempre, A veces, Casi<br>(Marque una en cada u | | | | | | | | - | kilos | | |
| | (Marque and en cada a | ina ae ias c | pres | juntusj | | | | | | | | |
| | <ol> <li>a. Nervioso/a? Diría</li> </ol> | I | | | | | Ah | ora | voy a k | eerle unas frases que q | uizás s | ean ciertas o no |
| | □ Siempre | | | Casi | nunc | a | en | cua | anto a e | ste parque. | | |
| | □ Casi siempre | 2 | | Nun | a | | | | | | | |
| | ☐ A veces | | | | | | | | | | | |
| | | | | | | | 37 | . Pa | ara cada | a una de las frases, por | favor o | lígame si está |
| | b. Sin esperanza? Di | iría | | | | | | to | talmen | te de acuerdo, de acue<br>te en desacuerdo. | | |
| | □ Siempre | | | Casi | nunc | a | | | | | | |
| | □ Casi siempre | 2 | | Nun | a | | | | | | | |
| | □ A veces | | | | | | - | | | | | |

| | a. | Las personas de por aquí están dispuestas a ayudar a sus vecinos. Totalmente de acuerdo De acuerdo Ni de acuerdo ni en desacuerdo En desacuerdo Totalmente en desacuerdo | c. Se armó una pelea en el parque Muy probable Probable Ni probable ni improbable Improbable Muy improbable |
|---|---|---|---|
| | b. | Las personas que frecuentan este parque son de<br>confiar. | |
| | | ☐ Totalmente de acuerdo | PARA QUE EL ENTREVISTADOR LEA: Estamos pensando en |
| | | ☐ De acuerdo | desarrollar unos nuevos programas para la comunidad y las<br>siguientes preguntas solicitan su aportación sobre estos |
| | | ☐ Ni de acuerdo ni en desacuerdo | programas. |
| | | ☐ En desacuerdo | programas. |
| | | ☐ Totalmente en desacuerdo | |
| | c. | Las personas que frecuentan este parque por lo general no se llevan bien los unos con los otros. □ Totalmente de acuerdo | 39. Si pudiera recibir un premio pequeño por ir al parque,<br>¿cuál preferiría? |
| | | ☐ De acuerdo | ☐ Una botella para el agua |
| | | □ Ni de acuerdo ni en desacuerdo | Un protector labial |
| | | □ En desacuerdo | □ Una pelota |
| | | ☐ Totalmente en desacuerdo | ☐ Un frisbee |
| | | | ☐ Una tarjeta de regalo de iTunes<br>☐ Otra |
| | d. | Las personas que frecuentan este parque no | |
| | | comparten los mismos valores. | |
| | | ☐ Totalmente de acuerdo | 40. Si el premio fuera un boleto para la rifa de un artículo |
| | | □ De acuerdo | más grande, ¿qué premio le gustaría ganar? |
| | | □ Ni de acuerdo ni en desacuerdo | □ Un iPod |
| | | ☐ En desacuerdo | <ul> <li>Una computadora portátil tipo tableta</li> </ul> |
| | | ☐ Totalmente en desacuerdo | ☐ Un tarjeta de regalo de \$200 |
| | | | □ Otra |
| 38. | favo<br>imp | cada una de las siguientes frases, por favor dígame<br>or si es Muy probable, Probable, Improbable o Muy<br>robable que las personas en este parque hicieran las<br>ientes cosas | 41. ¿En qué clases de ejercicio participaría si se ofrecieran en este parque? (Marque todas las que correspondan) □ Aeróbicos □ Acondicionamiento físico |
| | Pers | onas en el parque hicieran algo si: | |
| | | | ☐ Baile hip hop ☐ Baile en línea |
| | a. | Algunos niños estuvieran pintando o escribiendo | ☐ Kickboxing o boxeo tailandés |
| | | con aerosol (grafiti) | □ Pilates |
| | | ☐ Muy probable | □ Salsa |
| | | □ Probable | ☐ Club para caminar |
| | | □ Ni probable ni improbable | ☐ Yoga |
| | | □ Improbable | ☐ Zumba |
| | | ☐ Muy improbable | □ Otra |

.

| 42. | | ante la semana, ¿cuál sería la mejor hora para que<br>d participara en estas clases? | 44. ¿Tiene comentarios adicionales sobre este parque? |
|---|---|---|---|
| | | La mañana (de las 7 a las 10) | |
| | | Las horas del mediodía (de las 10 a la 1) | |
| | | La tarde (de la 1 a las 5) | |
| | | El comienzo de la noche (de las 5 a las 8) | |
| | | La noche (después de las 8) | |
| 43. | | ante el fin de semana, ¿cuál sería la mejor hora para<br>usted participara en estas clases? | |
| | | La mañana (de las 7 a las 10) | Este es el final del cuestionario. |
| | | Las horas del mediodía (de las 10 a la 1) | Muchas gracias por su participación. |
| | | La tarde (de la 1 a las 5) | |
| | | El comienzo de la noche (de las 5 a las 8) | |
| | | La noche (después de las 8) | l |
| 45. | Desp | oués de terminar la encuesta, entre la letra (A – J) que co | orresponde al tipo de constitución física del entrevistado. |
| | _ | (Entra una letra A – J) | |

# Appendix E: Body type categories



#### Appendix F: Park user interview recruitment guide

# **Park User Sample**

*Interview only those over age 18.* No exceptions! Before conducting an interview, verify the age of the person. You are *not* permitted to speak to children even if a parent is present!

If the park is busy during a given shift, try to conduct additional surveys. However, conducting additional interviews on one day does not reduce the number of interviews required for the next day.

Try to interview people that are representative of the people using the park on any given day. Take into consideration activity level (active/sedentary), gender (men/women), and race.

## **Survey Introduction**

When inviting perspective participants to answer the survey, explain that you are working with AltaMed and the RAND Corporation to evaluate how well the parks are serving the local community. Explain that getting opinions from Park Users is critical. Tell prospective participants that the questionnaire will take only a few minutes of their time, and that the results will be given to the Department of Recreation and Parks to help improve local parks. When requested, give interviewees a flyer, which explains more about the project.

# **Selecting Participants**

Park users will be selected using a quota design, meaning that you will need to interview a certain number of people according to their characteristics, such as gender and activity level.

- 1. In each park, interview 15 females and 15 males
- 2. For each gender interview 3-5 people who have just been engaging in some physical activity, the remainder will be individuals who are sedentary. In other words, you will interview 5 active males, and 10 sedentary males, 5 active females, and 10 sedentary females.
- 3. Participants can be recruited from any target area with people in it.
  - a. You may choose to start on any point in the target area (i.e., you do not have to start on the left side). After attempting to recruit the first participant, walk through the target area such that you cover the whole target area without repeating any part of it. For example, start in one corner and move clockwise around the area, or counter-clockwise.
  - b. As you walk through the target area, attempt to recruit every other person that you encounter.
  - c. Once you have covered the entire target area as explained above, move to another target area with people in it.
- 4. Avoid concentrating on a single age group (e.g., all seniors).
- 5. There are no special instructions related to the race/ethnicity of participants. However, note that in some parks you should expect to interview more individuals of certain race/ethnicity groups.
  - a. Poinsettia RC and Hoover RC, expect to interview more White participants.
  - b. St. Andrews RC, Van Ness RC, Jim Gilliam RC, expect to interview more Black participants.
  - c. Alpine RC and Seoul International RC, expect to interview more Asian participants.
  - d. In all other places, expect to interview a majority of Latino participants.

# Administration

On each survey there are two required fields to help track adherence to the quota design: 1) Gender, and 2) Activity level. These fields must be completed before proceeding to the rest of the survey questions.

#### Appendix G: Household interview recruitment guide

## **Household Sample**

Interviewers will survey residents living at designated addresses within one quarter (1/4 mile), one half (1/2 mile), and one (1 mile), of the park. RAND will identify residential addresses within each of these three different distance areas and provide them to Interviewers by the first day of each park observation. The goal is to interview members of 10 households in each stratum, or complete 30 interviews.

The Interviewer (you) will need to determine if those addresses are appropriate for including in the study. In some cases, multiple residences may be associated with a single address (e.g. apartment buildings) or the address may not be valid (e.g., commercial buildings, vacant lots, condemned home). You must follow the established protocols to ensure that the interviewing methods meet scientific research criteria.

#### **Selecting Apartments**

When the provided address is to an apartment building, individual units are determined as follows:

- 1. The **1**<sup>st</sup> **time** you encounter this scenario, take the stairs to the **second floor** of the building. Approach the **first apartment to the right.** This protocol should be followed for all oddly numbered subsequent occurrences (3<sup>rd</sup> time, 5<sup>th</sup> time, 7<sup>th</sup> time, etc.). [If the apartment building is a single story, follow the directions in #2.]
  - a. On the Household Interview Log, enter the apartment number next to the printed address AND note that the apartment is on the second floor.
- 2. The **2**<sup>nd</sup> **time** you encounter this scenario, select the **first apartment to the right** on the **first floor** of the building. This protocol should be followed for all evenly numbered subsequent occurrences (2<sup>nd</sup> time, 4<sup>th</sup> time, 6<sup>th</sup> time, etc.).
  - a. On the Household Interview Log, enter apartment number next to the printed address AND note that the apartment is on the first floor.

#### **Selecting Freestanding Units**

When there is more than one freestanding unit at the provided address, determine which unit to approach as follows:

- 1. The **1**<sup>st</sup> **time** you encounter this scenario, select the **first unit** you approach when walking onto the property. This protocol should be followed for all oddly numbered subsequent occurrences (3<sup>rd</sup> time, 5<sup>th</sup> time, 7<sup>th</sup> time, etc.).
  - a. On the Household Interview Log, enter the unit number (e.g., Unit A or front house) next to the printed address.
- 2. The **2**<sup>nd</sup> **time** you encounter this scenario, select the **second unit** you approach when walking onto the property. This protocol should be followed for all evenly numbered subsequent occurrences (2<sup>nd</sup> time, 4<sup>th</sup> time, 6<sup>th</sup> time, etc.).
  - a. On the Household Interview Log, enter the unit number (e.g., Unit B or back house) next to the printed address.

#### Selecting Alternative Addresses

It is important that you attempt an interview at each address on the list. If, however, an address is invalid or a residence is not occupied (e.g., a condemned building or vacant lot), select an alternative residence as follows:

- 1. Replace a **single-family residence** by identifying the property located to the immediate **left** of the original address. [If there is more than one residence at the identified address (e.g., apartment), skip to Action #2.]
  - a. If the property to the left is a **single-family residence**, note the replacement address under the "Alternative Address" column on the Household Interview Log. It is also necessary to indicate whey the alternative address was selected under the "Reason For Alternative Address" column on the log.
  - b. If the building to the left is an **apartment building or multiple freestanding units** follow the protocol outlined in the *Selecting Apartments* and *Selecting Free-Standing Units*. Note the replacement address under the "Replacement address" column on the Household Interview Log. It is also necessary to indicate why an alternative address was selected under the "Reason for replacement" column on the log.
  - c. If there is a **vacant lot or commercial building** to the left of the original address, continue to search for a residential property as follows:
    - Continue walking to the left of the original address. If you come to the end
      of the street without identifying an appropriate replacement address,
      return to the original address and follow the same protocol by walking to
      the right.
    - ii. If you come to the end of the street without identifying an appropriate replacement address, return to the original address. Then follow the same protocol starting at the address located immediately across the street (first walking right and then left, if necessary).
      - If no residential replacements are identified, note this on the Household Interview Log by writing "no replacement located" under the "Replacement address" column. If, however, a replacement address was determined, indicate the address on the log. It is also important to write in the reason for selecting an alternative address on the log.
- Replace an apartment by selecting the first occupied unit to the left of the original unit.
   This scenario only applies IF the apartment identified when following the protocol outlined in the Selecting Apartments section yields an unoccupied unit (no people are currently residing in the unit).
  - a. If you come to the end of a hallway, return to the original unit and continue searching for an occupied unit to the right. If there are no occupied apartments on the same floor as the original unit, select the next highest floor, and so on. If no occupied units are identified, note this on the Household Interview Log by writing "no replacement located" under the "Replacement address" column. If a replacement address was determined, indicate the unit and floor number on the log. It is also important to write in the reason for selecting an alternative address on the log.
- 3. Replace a freestanding unit by selecting the first occupied unit encountered while walking beyond the originally unit If no occupied units are identified, note this on the Household Interview Log by writing "no replacement located" under the "Replacement address" column. If a replacement address was determined, indicate the unit and floor number on the log. It is also important to write in the reason for selecting an alternative address on the log.

#### **Selecting Interview Participants**

When the appropriate residential address has been identified, knock on the door or ring the doorbell. When the door is answered, immediately explain who you are and why you are there. Proceed by asking to speak with the person who is **over 18**, **currently at home**, **with the next birthday**. Ask this person to participate in the interview process and notify her/himof the incentive. If this person declines, continue asking for participation until some agrees to participate or all people over the age of 18 refuse participation.

#### **Attempted Interviews**

Make a total of four attempts to interview a person at each selected address. When returning to an address, always approach the same door as your initial attempt (e.g., front door or same apartment number). If no one answers the door, note the date AND time (e.g., AM or PM) next to the appropriate attempt check box in the "Attempts" column on the Household Interview Log.

If a minor answers the door and indicates there is no one over the age of 18 available, indicate the date AND time (e.g., AM or PM) next to the appropriate attempt check box in the "Attempts" column on the Household Interview Log. In the same space, indicate that a child was home by writing "minor only" above the date and time.

# **Conducting Interviews**

For safety, always conduct surveys in the presence of another Interviewer. You should never enter a residence when talking with survey participants. Rather, conduct all interviews at the door. After you complete an interview, check the appropriate box in the "Outcome" column of the Household Interview Log to indicate that the person agreed to participate in the interview, and if it was conducted on the iPad or on a paper form. Note the date in the "Contact date" column.

Participants have the right to stop an interview at any time. If this happens, check the appropriate iPad or Paper box in the "Outcome" column and write "stopped" above the box that you checked in the "Outcome" column. Record the date as usual in the "Contact date" column.

#### Refusals

When residents (over age 18) indicate that they are unwilling to participate in the interview, note the refusal on the Household Interview Log by circling "Refusal" in the "Outcome" column. The date should be noted under the "Contact date" column.

When residents decline to participate, DO NOT attempt to conduct another interview at this address. Choose a replacement address from the alternatives provided.

#### No Contact

Each time you attempt contact at a residence you should circle the appropriate number in the "Attempts" column. If no contact was made with a resident (at least 18 years of age) after four attempts, make sure that each of the numbers is circled, and write "No contact" in the "Contact date" column.

#### **Safety Considerations**

If you become concerned about your health and/or safety (e.g., drugs, violence, dogs) while attempting to conduct interviews, leave the area immediately. Make a notation on the Household Interview Log to indicate the situation (e.g., Stopped due to safety). When possible, select an alternative address as a replacement.

# Appendix H: Oral consent script

# Promoting Physical Activity in High Poverty Neighborhoods Oral Consent Script

| Hi, |
|---|
| I am and I work with AltaMed Health Services and the RAND Corporation. In association with the LA City Department of Recreation and Parks we are conducting research funded by the National Institutes of Health to try to learn more about how people use the parks and how we can improve them. Would you mind participating in a brief survey that will take about 10-15 minutes? I can offer you a (incentive type) as a token of appreciation for your time. Your participation is anonymous and voluntary you can choose to stop at any time. We don't need to know your name. I have a brief description of the study if you want more information and a number you can call and if you have any questions. Are you willing to participate?" |
| Are you 18 or over? |
| (If NO, stop) |
| (If YES, proceed) |
| PROMOTING PHYSICAL ACTIVITY IN HIGH POVERTY NEIGHBORHOODS |
| Guión para la obtención verbal del consentimiento |
| Hola: |
| Me llamo y trabajo con AltaMed Health Services y con RAND Corporation. En conjunto con el Departamento de Recreación y Parques de la ciudad de Los Ángeles estamos realizando una investigación financiada por los Institutos Nacionales de Salud para averiguar más acerca de cómo usan las personas los parques y cómo podemos mejorarlos. ¿Le importaría participar en una encuesta breve que dura entre 10 y 15 minutos? Puedo ofrecerle un(a) (un obsequio) en agradecimiento por el tiempo que nos dedique. Su participación es anónima y voluntaria. Puede dejar de participar en cualquier momento. No necesitamos saber su nombre. Si desea más información, tengo una descripción breve del estudio. También tengo un número telefónico al que puede llamar si tiene preguntas. ¿Está dispuesto(a) a participar? |
| ¿Tiene 18 años o más? |
| (Si la respuesta es "No", pare aquí) |
| (Si la respuesta es "Sí", continúe). |

# Appendix I: Project summary (English and Spanish)



#### **NEIGHBORHOOD PARKS**

**Neighborhood Parks** is a project which has the goal is of finding out the best way to help people in the City of Los Angeles become more physically active in their local parks. The Project will begin in June, 2013, and we will invite selected park users and local residents like you to participate in an interview on this topic. We will ask about your park use, your health, and your opinions about park programs.

In addition to interviews, members of our Project team will visit your local park on randomly selected days and times in order to see how many people are there and how active they are.

Once we find out what you think about the parks and how often they are being used, we will then create new programs to encourage more people to be active in the park. These will include free classes and a "loyalty" program, where people can earn rewards for visiting the park frequently. After we launch the programs, we will return to the parks to interview more people and see if the programs worked.

**Neighborhood Parks** is a joint effort between The City of Los Angeles Department of Recreation and Parks, AltaMed (a healthcare service provider) and The RAND Corporation, a private, non-profit organization that conducts research and analysis to help improve public policy and decision-making.

**Neighborhood Parks** is funded by the National Heart, Lung, and Blood Institute (NHLBI) of the National Institutes of Health (NIH).

# Questions?

- Contact Project Director Terry Marsh, (310) 393-0411 ext.
   6846
- The Principal Investigator of the study is Dr. Deborah Cohen, (310) 393-0411 ext. 6023
- The contact for RAND's Human Subjects Protection Committee is James Tebow, (310) 393-0411, ext. 7173



#### **PARQUES DE VECINDARIO**

**Parques de vecindario** es un proyecto cuyo objetivo es averiguar la mejor forma de ayudarles a los habitantes de la ciudad de Los Ángeles a realizar más actividad física en los parques cercanos a su lugar de domicilio. El proyecto comenzará en junio de 2013. Invitaremos a usuarios seleccionados de los parques y a residentes de la zona como usted a participar en una entrevista sobre este tema. Le haremos preguntas sobre el uso del parque, sobre su salud y sobre sus opiniones acerca de los programas del parque.

Además de hacer las entrevistas, los miembros del equipo del proyecto visitarán el parque de su localidad a distintas horas en distintos días para ver cuántas personas hay allí y qué tan activas son.

Cuando averigüemos lo que usted opina acerca de los parques y veamos con qué frecuencia los usa la comunidad, crearemos nuevos programas que estimulen a más personas a realizar actividad física allí. Entre ellos se cuentan clases gratuitas y un programa de «usuario leal y frecuente» en el que las personas pueden ganar premios por visitar el parque a menudo. Después del lanzamiento de los programas, regresaremos a los parques a entrevistar a más personas y ver si los programas funcionaron.

Parques de vecindario es una iniciativa conjunta del Departamento de Recreación y Parques de la ciudad de Los Ángeles, AltaMed (una compañía que proporciona atención médica) y RAND Corporation (una organización privada sin fines de lucro que realiza investigaciones y análisis a fin de mejorar las políticas públicas y la toma de decisiones).

El proyecto cuenta con financiación del Instituto del Corazón, los Pulmones y la Sangre (NHLBI, por sus siglas en inglés), que forma parte de los Institutos Nacionales de Salud (NIH).



# ¿Tiene preguntas?

- Comuníquese con Terry Marsh, director del proyecto, teléfono (310) 393-0411, ext. 6846
- Dra. Deborah Cohen es la investigadora principal del estudio, teléfono (310) 393-0411, ext.
   6023
- James Tebow es el contacto del comité de protección de sujetos humanos en investigaciones de RAND, teléfono (310) 393-0411, ext. 7173

# **EMERGENCY SERVICES**

**If you** or someone you know needs immediate mental health assistance or has a question about a mental health issue, we encourage you to **contact:** 

Los Angeles County Department of Mental Health Access Center 24/7 Helpline at:

1-800-854-7771

TYY for Hearing Impaired 562-651-2549

# **SERVICIOS DE EMERGENCIAS**

Si usted o alguien que conozca necesitan ayuda inmediata de salud mental o tiene alguna pregunta sobre un problema de salud mental, por favor llame a:

Departamento de Salud Mental Centro de Acceso de Los Ángeles línea de ayuda 24/7:

1-800-854-7771

Número para personas con deficiencias auditivas 562-651-2549

#### Appendix K: Data and safety monitoring plan

# Promoting Physical Activity in High Poverty Neighborhoods (HSPC Study ID: 2011-0692)

# **Data and Safety Monitoring Board**

We have created a study DSMB that is external to the project staff to review all protocols and interim findings, including questionnaires, recruitment progress, interim data findings, and data quality. The DSMB will be composed of a statistician (Bonnie Ghosh-Dastidar, RAND), an expert in physical activity (Dr. John Elder, professor at San Diego State University) and an expert in parks and physical activity (Dr. Myron Floyd, North Carolina State University).

The DSMB will monitor the overall conduct of the RCT and will ensure the overall safety of participants by protecting participants from avoidable harm and declaring clear benefit when there is proof beyond a reasonable doubt. The DSMB will meet at least once per year (or more as needed) by teleconference. If there are any adverse findings related to park improvements, these will be reported to the DSMB, our community partners (the Los Angeles Department of Recreation and Park, AltaMed Health Services), and the RAND HSPC. In addition, the DSMB will evaluate any adverse events (along with the HSPC) to protect the safety of study participants and study staff.

# **Data Monitoring Plan**

#### Data Collection and Management

All data collected will not have any personal identifiers. Randomization is at the park level, rather than the person level. All datasets will be password-protected.

Quality control procedures will utilized to ensure that park observations and recruitment is on schedule, treatment allocation is occurring as planned, data collection protocols are being used accurately.

A new quality control measure we would like to introduce is to take a photograph at one park target area during every observation. The photo will be time stamped and delivered with the data to RAND. Once received at RAND it will be deleted from the iPad mini. RAND staff will review the photo to validate the park user counts in that target area. Once it is reviewed by RAND, it will be stored in password protected file and will be deleted at the end of the study. It will be coded with the date, park ID number, and park target area.

#### Data Storage

Data will be collected by AltaMed Promotoras (field staff) on password protected iPad minis and will be uploaded to Accellion. Computer files will be password protected with restricted access to project staff. All analytic data files and databases will be maintained on a secure, password-protected server. iPad minis will be have a password protected ID known only to team members.

# Data Transfer

Electronic data will be transferred from the iPad mini to RAND via Accellion. The data include the park observational data as well as the survey data (which do not contain any personal identifiers).

# **Elements of Safety Monitoring Plan**

Reporting of Adverse Events

For this study, we will define an adverse event (AE) as any untoward physical or mental health occurrence that may present itself during the conduct of the study and that may or may not have a causal relationship with the study procedures.

For the baseline measurement, our greatest concern is the safety of the study staff that will be visiting parks in low income neighborhoods in pairs. They are trained to be careful and never to approach any person who appears intoxicated or mentally ill. If they see any illegal activity, such as drug deals, they are advised to leave the scene immediately. They are to carry cell phones and wear comfortable shoes.

We will use the FDA definition of serious adverse event (SAE), which is any adverse experience occurring during the intervention that results in any of the following outcomes: death, a lifethreatening adverse experience, or a persistent or significant disability/incapacity.

#### **Anticipated Adverse Events**

1. Suicidal ideation or intent to harm self

Field Interviewers will not be probing for this information, since it is not part of the research task. However, if a study respondent spontaneously reports immediate intent to commit suicide, field interviews will follow procedures below:

Emergency – In the rare instance that a respondent is in imminent danger and needs emergency medical or mental health services, the Field Interviewer will insure her own safety and then will dial 911 on her cell phone and request assistance. If a respondent reports that they are thinking of committing suicide and has a plan to do so and then terminates the interview immediately after providing this information, this circumstance should be considered an emergency and the interviewer should dial 911 to request assistance. The Field Interviewer will immediately call the Project Coordinator and write and submit an incident report the same day.

The Project Coordinator will send an incident report to the RAND HSPC on the same day.

The Project Coordinator will consult with the RAND HSPC to determine whether further follow-up is needed.

Non-emergency —If a respondent spontaneously indicates that he/she is *thinking* about committing suicide (but has no immediate plan), the Field Interviewer will say:

"You seem to be having a difficult time. If you think this is an emergency, you can call 911 or another local emergency number such as the Mental Health Crisis Care [give 800 number]. If you think you need help with this problem, you can talk to your doctor, your therapist/counselor, or call a doctor/therapist in your area."

The Field Interviewer will also provide the respondent with a written list of mental health referral numbers and suggest that he or she discuss feelings with their regular physician or with a mental health specialist obtained through referral. The Field Interviewer will call the Project Coordinator within one hour after the interview. The Field Interviewer will complete an incident report the same day.

The Project Coordinator will send the incident report to the RAND HSPC within 24 hours.

The Project Coordinator will consult with the RAND HSPC to determine whether further follow-up is needed.

#### 2. Severe depression

The new survey instrument includes some questions about mental health. If the respondent appears to get very upset by these questions (either during or after the interview) and/or spontaneously discloses that they feel very depressed, the Field Interviewer will say:

"You seem to be having a difficult time. If you think this is an emergency, you can call 911 or another local emergency number such as the Mental Health Crisis Care [give 800 number]. If you think you need help with this problem, you can talk to your doctor, your therapist/counselor, or call a doctor/therapist in your area."

The Field Interviewer will also provide the respondent with a written list of mental health referral numbers and suggest that he or she discuss feelings with their regular physician or with a mental health specialist obtained through referral. The Field Interviewer will call the Project Coordinator within one hour after the interview. The Field Interviewer will complete an incident report the same day.

# 3. Serious injury during physical activity class

Part of the intervention involves offering additional physical activity classes at select parks. We will be working closely with Park Directors in implementing these classes.

In addition, all activity instructors will administer verbal consent for participation in exercise classes in the parks, specifying that if potential participants have health concerns, of if they are over 60 and have never exercised before, they should talk to their doctor before participating in the classes.

All Activity Instructors will be trained on park procedures regarding in how to respond in the event that someone is injured or otherwise needs medical attention while participating in class. These include:

<u>Emergency</u> – In the rare instance that a respondent is in imminent danger and needs emergency medical services, the Activity Instructor will dial 911 on his or her cell phone and request assistance. The Instructor will also notify the Park Director (or park staff in charge if the Director is not there) and will notify the Project Coordinator and write and submit an incident report the same day.

The Project Coordinator will send an incident report to the RAND HSPC on the same day.

The Project Coordinator will consult with the RAND HSPC to determine whether further follow-up is needed.

<u>Non-emergency</u> – If a respondent is injured or becomes ill, but it is not an emergency, Activity Instructors will contact the Park Director (or park staff in charge if the Director is not there) and will notify the Project Coordinator and write and submit an incident report the same day.

The Project Coordinator will send the incident report to the RAND HSPC within 24 hours.

The Project Coordinator will consult with the RAND HSPC to determine whether further follow-up is needed.

# Appendix L: Data Log

Two data logs will be used in each park (or four during reliability data collection periods). The first page (Parks Data Log) summarizes data collection to date, while the second (Park User Interview Log) and subsequent pages are used to record daily park user interviews.

| | PARKS DATA LOG |
|-------|----------------|
| Park: | |

| Name | Date & Day of week | Park int | erviews | Household | interviews | Station interviews | |
|---|---|---|---|---|---|---|---|
| Name | Date & Day of Week | iPad | Paper | iPad | Paper | iPad | Paper |
| | Sub-total | | | | | | |
| | TOTALS | | | | | | |

| User |
|------|

| | Park n | ame: | | Date: | | | |
|---|---|---|---|---|---|---|---|
| Pro | motora n | ame: | | | | | |
| # | Target<br>Area | Gender<br>M = Male<br>F = Female | Race/Ethnicity L = Latino B = Black W = White O = Other | Age Group<br>Ad = Adult<br>Sr = Senior | Activity Level<br>S = Sedentary<br>A = Active | Outcome<br>I = iPad<br>P = Paper<br>R = Refuse | Comments |
| 1 | | M F | L B W O | Ad Sr | S A | I P R | |
| 2 | | M F | L B W O | Ad Sr | S A | I P R | |
| 3 | | M F | L B W O | Ad Sr | S A | I P R | |
| 4 | | M F | L B W O | Ad Sr | S A | I P R | |
| 5 | | M F | L B W O | Ad Sr | S A | I P R | |
| 6 | | M F | L B W O | Ad Sr | S A | I P R | |
| 7 | | M F | L B W O | Ad Sr | S A | I P R | |
| 8 | | M F | L B W O | Ad Sr | S A | I P R | |
| 9 | | M F | L B W O | Ad Sr | S A | I P R | |
| 10 | | M F | L B W O | Ad Sr | S A | I P R | |
| 11 | | M F | L B W O | Ad Sr | S A | I P R | |
| 12 | | M F | L B W O | Ad Sr | S A | I P R | |
| 13 | | M F | L B W O | Ad Sr | S A | I P R | |
| 14 | | M F | L B W O | Ad Sr | S A | I P R | |
| 15 | | M F | L B W O | Ad Sr | S A | I P R | |

At the end of the day, record the number of park user interviews completed in each category. Add the sub-total from the preceding day to your daily total, and enter the sum in the appropriate sub-total box.

| | Fen | nale | Male | |
|-------------|-----------|--------|-----------|--------|
| | Sedentary | Active | Sedentary | Active |
| Daily total | | | | |
| Sub-total | | | | |

Note that this page is to be duplicated for each day of data collection (i.e., each data collector should complete one of these pages for each day of data collection in every park. A single packet can be made with one Parks Data Log followed by six park user interview logs (possibly more for makeup days).

# Appendix M: Setting the network IP address

The instructions below explain how to set the IP address for the Rand Wireless network. Only RAND staff who have admin rights on the field laptop are permitted to make these changes. The intent is to have Rand Wireless be set as a static IP. However, if the laptop is connected to a network other than Rand Wireless, the steps listed below may have to be repeated in order to reestablish the network.

1. Open the Start menu and type cmd in the Search box and press enter.



2. Type ipconfig/all and press enter.

```
C:\Windows\system32\cmd.exe

Microsoft Windows (Version 6.1.76011
Copyright (c) 2009 Microsoft Corporation. All rights reserved.

C:\Users\lraaen>ipconfig/all
```

3. Scroll down until you see the DNS Servers and note what they are.

4. Open the Network and Sharing Center



5. Click on Change Adapter Settings.



6. Right click on the Rand Wireless connection and then click on Properties. Enter Admin username and password.



1.

2.

3. Select Internet Protocol Version 4 (TCP/IPv4) and click OK.



4. Click on the Use the following IP address button. Enter the preferred IP address (192.168.1.5), Subnet mask (255.255.255.0), Default gateway (192.168.1.1), and DNS server. Click OK.

